CLINICAL TRIAL: NCT02825563
Title: Phase I Additional Study of Anlotinib on Pharmacokinetics to Assess the Effect of High Fat Diet in Advanced Cancer Patients
Brief Title: A Phase I Study of Anlotinib on Pharmacokinetics to Assess the Effect of High Fat Diet in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-I-05
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anlotinib(In the fasting state) (Experimental): In the fasting state, Anlotinib po only once and after 14 days it could be continued by Qd po.until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Anlotinib(In the high fat diet state) (Experimental): In the high fat diet state, Anlotinib po only once and after 14 days it could be continued by Qd po.until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — in the fasting state
  Arms: Anlotinib(In the fasting state)
Drug: Anlotinib — in the high fat diet
  Arms: Anlotinib(In the high fat diet state)

SUMMARY:
The purpose of this study is to further study the pharmacokinetic characteristics of Anlotinib in Advanced Cancer Patients with High Fat Diet.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Advanced solid tumors( Non-small Cell Lung Cancer.Soft Tissue SarcomaMedullary. Thyroid Carcinoma)
* At least one measurable lesion (by RECIST1.1)
* Lack of the standard treatment or treatment failure
* 20≤BMI≤25
* 18-70 years,ECOG PS:0-1,Life expectancy of more than 3 months
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Clear allergies to the study drug or its ingredients
* Had the disease to affect drug absorption and metabolism
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Brain metastases patients with symptoms or symptoms controlled < 1 months
* Used any drugs inhibit or induce hepatic drug metabolic enzymes in 30 days before the study
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* Patients participated in other anticancer drug clinical trials within 4 weeks
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Anlotinib (in whole blood):Peak Plasma Concentration(Cmax) | up to 14 Days
  Peak Plasma Concentration(Cmax),Cmax in ng/mL.In the study , full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H96/H144/H192/H240/H336(H mans Hour).
Pharmacokinetics of Anlotinib (in whole blood):Area under the plasma concentration versus time curve (AUC) | up to 14 Days
  Area under the plasma concentration versus time curve (AUC), AUC in ng.h/mL.In the study , full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H96/H144/H192/H240/H336(H mans Hour).

SECONDARY OUTCOMES:
Pharmacokinetics of Anlotinib (in whole blood):Peak time（Tmax） | up to 14 Days
  Peak time（Tmax）,Tmax in h.In the study , full PK profiles will be obtained at H0/H1/H2/H4/H8/H11/H24/H48/H96/H144/H192/H240/H336(H mans Hour).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided